CLINICAL TRIAL: NCT02832596
Title: Changes in Measured Plasma Volume, Glycocalyx and Atrial Natriuretic Peptide During Anaesthesia, a Randomised Clinical Trial
Brief Title: Changes in Measured Plasma Volume, Glycocalyx and Atrial Natriuretic Peptide During Anaesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Tor Damén, Doctor, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Plasmavolume TDamen
Record Dates: First submitted 2016-07-11; First posted 2016-07-14 (Estimated); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Blood Pressure; Anesthesia
Keywords: Anesthesia; Blood pressure; Plasma Volume; Vasopressor agents; Coronary artery bypass; Glycocalyx; ANP; Coagulation
MeSH Terms: conditions — Thrombosis | interventions — Norepinephrine; Vasoconstrictor Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Ordinary anesthesia, mean arterial pressure allowed to decrease to 60 mmHg. If it is lower the patients will receive a norepinephrine infusion in order to raise the mean arterial pressure to 60 mmHg.
- Maintained blood pressure (Active Comparator): Ordinary anaesthesia and maintained preanesthetic blood pressure by norepinephrine infusion
  Interventions: Drug: Norepinephrine; Procedure: Maintained blood pressure

INTERVENTIONS:
Drug: Norepinephrine — Ordinary anaesthesia and maintained preanesthetic blood pressure by norepinephrine infusion
  Other Names: Vasopressor
  Arms: Maintained blood pressure
Procedure: Maintained blood pressure — Norepinephrine therapy to maintain preanesthesia blood pressure
  Arms: Maintained blood pressure

SUMMARY:
The arterial blood pressure is thought to affect the ratio between filtration and reabsorption of fluids in the circulating blood volume and thereby the plasma volume. During induction of anesthesia blood pressure, hemoglobin level and hematocrits decreases and the plasma volume increases. The aim of the study is to evaluate weather a maintained blood pressure with norepinephrine during anesthesia induction reduces the increase in 125 iodine-labeled human serum albumine (125I-HSA) measured plasma volume.

DETAILED DESCRIPTION:
24 patients scheduled for coronary artery bypass surgery will be included and randomized to receive either norepinephrine in the dose needed to maintain pre-anesthesia blood pressure or to a control group and receive norepinephrine only if mean arterial pressure decreases below 60 mmHg. Equal anesthesia in both groups will be monitored. No fluids will be infused.

Changes in vascular resistance and cardiac output will be measured with thermodilution and changes in plasma volume will be measured with 125I-HSA.

Endothelial cell function will be evaluated by measuring leakage of 125I-HSA and the plasma concentration of endothelial cell markers. Hormonal effects will be evaluated by measuring the plasma concentration of atrial natriuretic peptide (ANP). Shedding of glycocalyx will be evaluated by measuring heparan sulphate. The level of fibrinogen and platelet function will be evaluated by thromboelastography/multiplate.

ELIGIBILITY:
Inclusion Criteria:

* Elective coronary artery surgery patients

Exclusion Criteria:

* Age under 40 years
* Untreated hypertension
* A reduced left ventricular systolic ejection fraction of 45% or less
* Diabetes mellitus
* Former stroke and/or a known carotid artery stenosis

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-10; Primary Completion 2019-08-20 (Actual); Study Completion 2019-08-20 (Actual)

PRIMARY OUTCOMES:
The change of plasma volume measured by 125I-HSA before anesthesia induction until 50 minutes after anesthesia induction. | 50 minutes from anesthesia induction
  To assess if the increase in plasma volume measured by 125I-HSA can be reduced by maintaining the blood pressure with vasopressor infusion.

SECONDARY OUTCOMES:
Difference in 125I-HSA leakage | 50 minutes from anesthesia induction
  To assess if there is a difference in 125I-HSA leakage in between the control and intervention groups before and after anaesthesia induction
ANP, heparan sulphate, thrombomodulin, fibrinogen, ROTEM | 50 minutes from anesthesia induction
  To assess if there is a difference in the plasma concentration of ANP, heparan sulphate, thrombomodulin, fibrinogen and ROTEM before and after anaesthesia induction in the intervention group compared to the control group

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Nygren, MD PHD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided